CLINICAL TRIAL: NCT00227487
Title: The Evaluation of Intestinal Inflammation and Carbohydrate Digestion in Children With Autistic Spectrum Disorders
Brief Title: Intestinal Inflammation and Carbohydrate Digestion in Autistic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Rafail Kushak, Ph.D., Assistant in Biochemistry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KRPP1
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Autism; Inflammation
Keywords: autism; intestine; disaccharidases; inflammation; permeability
MeSH Terms: conditions — Autistic Disorder; Inflammation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stool collection, Carbohydrate administration, Questionnaires (Other): A stool sample will be obtained
  A carbohydrate solution (lactulose plus rhamnose dissolved in tap water) will be administered during a clinically indicated endoscopic procedure.
  Five questionnaires will be completed by parent/guardian
  Interventions: Other: Stool collection; Other: Administration of carbohydrate solution during clinically indicated endoscopy; Other: Questionnaires

INTERVENTIONS:
Other: Stool collection — Stool sample will be obtained by parent at home to prevent sample dilution during the cleanout
Other: Administration of carbohydrate solution during clinically indicated endoscopy — * A carbohydrate solution (lactulose + rhamnose dissolved in tap water) will be administered during the procedure (upper endoscopy) through a catheter directly into the duodenum to allow for intestinal permeability analysis.
  * Clinically indicated pinch biopsies will then be obtained.
  * The endoscopy procedures will take at least 1 - 1 ½ hours.
  * Children will then typically recover in the endoscopy suite for 2 - 2½ hours or less, if the child is medically cleared to leave the endoscopy suite sooner.
  * Urine for intestinal permeability analysis will be collected during 5 hours after carbohydrate solution administration. If the child has not voided, an additional 60 minutes will be allowed for the child to void. If the child is not continent for urine, a bag will be applied to catch the specimen.
Other: Questionnaires — Parents/legal guardians of subjects will be asked to complete five (5) questionnaires: the Gastrointestinal Symptoms Inventory; a Developmental Screening for Autism - based on the child's age, either the Checklist for Autism in Toddlers (CHAT), Modified Checklist for Autism in Toddlers (M-CHAT), or the Social Communication Questionnaire (SCQ); the Behavior and Sensory Interest Questionnaire (BSI), the Behavior Problems Inventory (BPI), and the Aberrant Behavior Checklist (ABC). It should take parents/guardians no longer than eighty-five (85) minutes to complete all 5 surveys. Results from these questionnaires will be correlated with documented gastrointestinal and/or neurological diagnostic information from subject medical records and with research study test results.

SUMMARY:
The purpose of the study is to find correlations between non-invasive fecal tests of intestinal inflammation and macro- and microscopic evaluation of duodenal and colonic histology, disaccharidase activity, and intestinal permeability in children with autism.

DETAILED DESCRIPTION:
Gastrointestinal disorders in children with autism receive little attention. However, symptoms such as abdominal pain, diarrhea, constipation, and flatulence have been considered contributing to the behavioral problems. These symptoms are associated partially with the deficiency of enzymes digesting carbohydrates and inflammation of the gastrointestinal tract. The effect of intestinal inflammation on neurological disorders experienced by autistic children remains unclear. We will study this problem using recently developed non-invasive tests based on two proteins (calprotectin and lactoferrin) analysis in children's stool. Activity of enzymes needed for carbohydrate digestion will be tested in small samples of intestinal tissue. Intestinal permeability will be assessed by measuring urinary excretion of carbohydrate substances (lactulose and rhamnose) administered via the endoscope. This test will help to determine if intestinal inflammation contributes to a "leaky" gut syndrome. The study will provide valuable information for understanding the association between gastrointestinal disease and behavioral problems in autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 months to 17 years inclusive.
* Subjects referred to a Massachusetts General Hospital for Children (MGH Main Campus or satellite clinic) for pediatric care or pediatric gastroenterology care.
* Subjects with documented gastrointestinal symptoms requiring endoscopy and duodenal pinch biopsy for disaccharidase activity evaluation for the standard medical treatment of gastrointestinal symptoms (i.e. endoscopy and biopsy cannot be performed solely for research purposes).

Exclusion Criteria

* Use of any proteolytic digestive enzyme supplements: prescription or over-the-counter (e.g., Pancrease [Creon-10], Lactase, etc.) up to 7 days prior to EGD with biopsy.
* Diagnosed bleeding disorder
* Hypoalbuminemia
* Unstable respiratory status evidenced by a diagnosed respiratory condition (such as asthma) that is not adequately controlled (e.g. evidence of repeated hospitalizations for exacerbations in asthma symptoms, etc.).
* Unstable cardiac status evidenced by a diagnosed cardiac condition.
* Nasal or menstrual bleeding. Additional blood in stool may effect calprotectin and lactoferrin concentration.

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2005-10; Primary Completion 2011-05 (Actual); Study Completion 2017-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Harland S. Winter, MD, Study Chair — Massachusets General Hospital; Timothy M Buie, M.D., Study Director — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

REFERENCES:
- [Derived] Kushak RI, Buie TM, Murray KF, Newburg DS, Chen C, Nestoridi E, Winter HS. Evaluation of Intestinal Function in Children With Autism and Gastrointestinal Symptoms. J Pediatr Gastroenterol Nutr. 2016 May;62(5):687-91. doi: 10.1097/MPG.0000000000001174. PMID 26913756
- See also: Related Info — http://www.partners.org